CLINICAL TRIAL: NCT03324191
Title: Effect of a Polyphenol-rich Tea Extract on Blood Lipid Response to Dietary Fat
Brief Title: Tea Extract, Blood Lipid and Dietary Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Lucozade Ribena Suntory (Industry)
Responsible Party: Principal Investigator, James Betts, Principle Investigator, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HVS-009
Record Dates: First submitted 2017-10-19; First posted 2017-10-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Lipid Metabolism; Diabetes
Keywords: Tea extract; Triglycerides; Energy metabolism
MeSH Terms: conditions — Diabetes Mellitus | interventions — Tea

STUDY DESIGN:
Intervention Model Description: Double-blind, single-centre randomised controlled trial using a cross-over experimental design.
Who Masked: Participant, Investigator
Masking Description: Participants and Researchers will be blinded to the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will consume 567 ml of plain water at least 1 hour before testing the trial.
  Information on dietary compliance will be collected. Participants will then be cannulated in an arm vein and a baseline fasting blood sample will be taken. Participants will be asked to consume a standard study meal challenge (providing 40 g dietary fat and less than 2 g carbohydrate or 1.2 g protein) and placebo drink within 15 min. Serial blood samples will be collected at baseline, 30, 60, 90, 120 and 180 min. The intervention will end once the 180 min sample is collected.
  For the tracer test subpopulation (n=15) the test meal will also contain 300 mg [1,1,1-13C3] tripalmitin to trace the incorporation of dietary lipid into plasma fatty acids.
  Interventions: Dietary Supplement: Placebo; Other: High fat liquid meal challenge
- Tea beverage (Experimental): Participants will consume 567 ml of plain water at least 1 hour before testing the trial.
  Information on dietary compliance will be collected. Participants will then be cannulated in an arm vein and a baseline fasting blood sample will be taken. Participants will be asked to consume a standard study meal challenge (providing 40 g dietary fat and less than 2 g carbohydrate or 1.2 g protein) and tea within 15 min. Serial blood samples will be collected at baseline, 30, 60, 90, 120 and 180 min. The intervention will end once the 180 min sample is collected.
  For the tracer test subpopulation (n=15) the test meal will also contain 300 mg [1,1,1-13C3] tripalmitin to trace the incorporation of dietary lipid into plasma fatty acids.
  Interventions: Dietary Supplement: Tea beverage; Other: High fat liquid meal challenge
- Tea extract (medium concentration) (Experimental): Participants will consume 567 ml of plain water at least 1 hour before testing the trial.
  Information on dietary compliance will be collected. Participants will then be cannulated in an arm vein and a baseline fasting blood sample will be taken. Participants will be asked to consume a standard study meal challenge (providing 40 g dietary fat and less than 2 g carbohydrate or 1.2 g protein) and concentrated tea extract at a medium concentration within 15 min. Serial blood samples will be collected at baseline, 30, 60, 90, 120 and 180 min. The intervention will end once the 180 min sample is collected.
  For the tracer test subpopulation (n=15) the test meal will also contain 300 mg [1,1,1-13C3] tripalmitin to trace the incorporation of dietary lipid into plasma fatty acids.
  Interventions: Dietary Supplement: Tea extract (medium concentration); Other: High fat liquid meal challenge
- Tea extract (high concentration) (Experimental): Participants will consume 567 ml of plain water at least 1 hour before testing the trial.
  Information on dietary compliance will be collected. Participants will then be cannulated in an arm vein and a baseline fasting blood sample will be taken. Participants will be asked to consume a standard study meal challenge (providing 40 g dietary fat and less than 2 g carbohydrate or 1.2 g protein) and concentrated tea extract at a high concentration within 15 min. Serial blood samples will be collected at baseline, 30, 60, 90, 120 and 180 min. The intervention will end once the 180 min sample is collected.
  For the tracer test subpopulation (n=15) the test meal will also contain 300 mg [1,1,1-13C3] tripalmitin to trace the incorporation of dietary lipid into plasma fatty acids.
  Interventions: Dietary Supplement: Tea extract (high concentration); Other: High fat liquid meal challenge

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo will be matched for flavour, odour, and colour, to a tea beverage, without any active ingredient (tea extract).
  Arms: Placebo
Dietary Supplement: Tea beverage — Tea beverage
  Arms: Tea beverage
Dietary Supplement: Tea extract (medium concentration) — Tea extract (medium concentration) will be matched for flavour, odour, and colour, to a tea beverage, with a medium concentration of tea extract.
  Arms: Tea extract (medium concentration)
Dietary Supplement: Tea extract (high concentration) — Tea extract (medium concentration) will be matched for flavour, odour, and colour, to a tea beverage, with a high concentration of tea extract.
  Arms: Tea extract (high concentration)
Other: High fat liquid meal challenge — A dairy based standard study meal challenge providing 40 g dietary fat and less than 2 g carbohydrate or 1.2 g protein.
  For the tracer test subpopulation (n=15) the test meal will also contain 300 mg [1,1,1-13C3] tripalmitin to trace the incorporation of dietary lipid into plasma fatty acids.

SUMMARY:
There are numerous factors known to determine the relative rate of lipid metabolism at rest between and within individuals, including: biological sex, endogenous carbohydrate availability, training status and, in particular, feeding. Recent focus has been placed on the potential of alternative nutrients, nutritional supplements and pharmacological agents to modify substrate selection in favour of greater lipid oxidation (e.g. caffeine, carnitine, green tea) and/or to alter lipid absorption (e.g. caffeine, carnitine, orlistat, green tea preparations).

Polyphenol-rich tea extract can have effects on lipase activity in the pancreas causing reduced fat absorption. The present study is to assess the potential for tea extract alone to be as effective at the liquid product in a western population.

DETAILED DESCRIPTION:
Participants will be asked to visit laboratories at the University of Bath on four occasions, with each visit separated by at least 2 days. Each visit will last approximately 5 hours.

Participants will be asked to provide informed consent to participate in the study and to answer a number of questions to confirm that it is safe for them to do so, and to confirm eligibility. Participants will be asked to monitor their diet for 48 h before their first laboratory visit, and then to replicate this diet before subsequent visits. Participants will also be asked abstain from caffeine (i.e tea and coffee), alcohol and strenuous physical activity the day before visiting us (e.g. no exercise that causing sweating or heavy breathing).

Participants will be asked to arrive to the laboratory after having not eaten for at least 5 hours, having drunk one pint of water at least one hour before testing. Upon arrival at the laboratory a person trained and experienced in sampling blood will insert a cannula (a small plastic tube) into a vein on the participants arm. This is to allow for repeated blood sampling every 30-60 minutes during their visit.

Participants will then be provided with one of the four supplements under investigation (i.e. either a placebo or one of the preparations derived from tea) to ingest as fluid along with a standard milkshake that provides participants with 40 g of fat, such that the appearance of this fat in the bloodstream can be measured. Of the 55 participants in this study, additional measurements will be made on a randomly selected sub-group of 15 to directly trace the appearance of fat in their blood samples; if participants have been asked and agreed to this part of the study then some of the fat in their milkshake would be a stable isotope tracer (13C-Tripalmitin). Participants will then rest comfortably, and a 10 ml sample of blood will be drawn from participants every 30 minutes for two hours, and at three hours, after consumption of the high fat drink.

ELIGIBILITY:
Inclusion Criteria:

1. Consent- Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
2. Age- Aged between 18 and 60 years.
3. Compliance- Understands and is willing, able and likely to comply with all study procedures and restrictions.
4. General Health - Good general and mental health with, in the opinion of the investigator or medically qualified designee:

   1. No clinically significant and relevant abnormalities of medical history or physical examination.
   2. Absence of any condition that would impact on the subject's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
5. No anticipated changes in diet and/or physical activity or lifestyle habits during the study period (e.g. pre-planned holidays, diets/exercise plan, smoking etc.)
6. Contraception- Females of childbearing potential who are, in the opinion of the investigator, practising a reliable method of contraception. Adequate contraception is defined as abstinence, oral contraceptive, either combined or progestogen alone OR injectable progestogen OR implants of levonorgestrel OR estrogenic vaginal ring OR percutaneous contraceptive patches OR intrauterine device or intrauterine system OR double barrier method (condom or occlusive cap [diaphragm or cervical vault caps] plus spermicidal agent [foam, gel, film, cream, suppository]) OR male partner sterilization prior to the female subject's entry into the study, and this male is the sole partner for that subject.

Exclusion Criteria:

1. Pregnancy- Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
2. Breast-feeding- Women who are breast-feeding.
3. Allergy/Intolerance- Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
4. Blood donation- More than 400ml of blood within 3 months of the screening visit and more than 1500ml of blood in the previous 12 months. Any reported bleeding disorder
5. Clinical Study/Experimental Medication

   1. Participation in another clinical study or receipt of an investigational drug within 90 days of the screening visit) to allow full recovery of blood volume
   2. Previous participation in this study.
6. Any reported recent (within 6 months) shift (>3 kg) in body mass
7. Substance abuse- Recent history (within the last 2 years) of alcohol or other substance abuse and / or Any reported use of substances which may pose undue personal risk to participants or introduce bias into the experiment as deemed by the Principal Investigator
8. Any reported condition or behaviour deemed by the Principal Investigator either to pose undue personal risk to the participant or introduce bias into the experiment
9. Exclusion criteria assessed after taking measurements- Those with body mass index < 18 or > 35 kg/m^2. Medical history of diabetes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Effect of tea extract on serum triacylglycerol concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls

SECONDARY OUTCOMES:
Effect of tea extract on systemic glucose concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic insulin concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic C-peptide concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic non-esterified fatty acid concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic high density lipoprotein concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic low density lipoprotein concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic glycerol concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic apolipoprotein A1 concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic apolipoprotein A2 concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic apolipoprotein B concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic apolipoprotein C2 concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic apolipoprotein C3 concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on systemic apolipoprotein E concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on plasma triacylglycerol concentration following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls
Effect of tea extract on the incorporation of dietary fats into systemic triacylglycerol following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls in a sub-population of 15 randomly selected participants.
Effect of tea extract on the incorporation of dietary fats into non-esterified fatty acids following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls in a sub-population of 15 randomly selected participants.
Effect of tea extract on whole body lipid oxidation following a high fat meal | 3 hour postprandial period
  Comparison of tea extract to placebo and positive controls in a sub-population of 15 randomly selected participants.

CONTACTS AND LOCATIONS:
Overall Officials: James Betts, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perkin OJ, Chen YC, Johnson DA, Thomas JE, Atkinson G, Betts JA, Gonzalez JT. Postprandial Metabolic Mesponses to High-fat Feeding in Healthy Adults Following Ingestion of Oolong Tea-Derived Polymerized Polyphenols: A Randomized, Double-blinded, Placebo-controlled Crossover Study. Am J Clin Nutr. 2023 Jul;118(1):132-140. doi: 10.1016/j.ajcnut.2023.04.020. Epub 2023 Apr 18. PMID 37080462